CLINICAL TRIAL: NCT07354295
Title: Multimodal AI-based Therapy Response Prediction and Risk Stratification for Esophageal Cancer
Brief Title: Integrating Multimodal AI to Predict Treatment Response and Refine Risk Stratification in Esophageal Cancer
Acronym: ECO
Status: Recruiting | Type: Observational
Sponsor: Shu Peng (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); Henan Provincial People's Hospital (Other); Zhongnan Hospital (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor-Investigator, Shu Peng, Dr, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 4059393
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; AI; prediction; prognosis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be obtained from residual specimens remaining after routine clinical laboratory testing, and tissue samples will be collected from specimens left over after pathologists have taken necessary sections for diagnostic purposes following surgical resection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Surgical resection cohort: neither neoajuvant therapy nor anti-tumor treatment prior to surgery
- neoadjuvant therapy cohort: received neoadjuvant therapy and esophagectomy
- conservative treatment: concervative treatment includes chemo/immuno/radiotherapy and targeted theray
- Endoscopic submucosal dissection (ESD): Endoscopic submucosal dissection (ESD)

SUMMARY:
This AI-driven model leverages multimodal data-such as radiomics, pathomics, genomics, and broader multi-omics profiles-to capture complementary aspects of tumor biology and predict treatment response and prognosis.

DETAILED DESCRIPTION:
Built upon retrospective cohorts for model development and rigorously validated in prospective cohorts, the proposed AI predictive model integrates multimodal data (radiomics, pathomics, genomics, and multi-omics)-each reflecting distinct dimensions of tumor heterogeneity-to enable joint prediction of treatment response and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically diagnosed esophageal cancer
2. Complete baseline clinical data available (including demographic characteristics, ECOG performance score, TNM staging, etc.)
3. No other primary malignant tumors
4. Provision of informed consent
5. Availability of pre-treatment CT imaging

Exclusion Criteria:

1. Imaging data quality insufficient for analysis
2. Presence of another primary malignant tumor
3. Severe systemic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with esophgeal cancer and have received treatment in Tongji hospital
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | From enrollment to the end of treatment at 3 years
  overall survival rate in 3-years

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Tongji medical college, Huazhong university of science and technology, Wuhan, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No
In accordance with the institution's data confidentiality requirements

REFERENCES:
- [Result] Xia T, Peng S, Yang F, Wang X, Yao W. Data-driven models in locally advanced oesophageal cancer. Lancet. 2025 Sep 27;406(10510):1334-1335. doi: 10.1016/S0140-6736(25)01766-0. No abstract available. PMID 41015514